CLINICAL TRIAL: NCT05850923
Title: The Efficacy of Speech Competition Training on Auditory Hallucination in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing SHI (Other)
Responsible Party: Sponsor-Investigator, Jing SHI, Nurse practitioner, Shanghai Mental Health Center
Organization: Shanghai Mental Health Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AH-IA-2021
Record Dates: First submitted 2023-04-19; First posted 2023-05-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Auditory Hallucination
Keywords: Schizophrenia; Intervention
MeSH Terms: conditions — Hallucinations; Schizophrenia

STUDY DESIGN:
Intervention Model Description: At first, all the participants will be randomized into a speech competition experimental group and a placebo control group, after 2 weeks the two interventions for two arms will be switch.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a speech competition experimental group (Experimental): The speech competition training was arranged twice a day, each lasting 15 minutes. The training included word search in sequence, word search out of order and word sorting. Patients need to follow the instructions in time for training. The reaction time, accuracy rate and the number of auditory hallucinations during the task were recorded.
  Interventions: Other: speech competition training
- Control group (Active Comparator): The patient will listen to the soothing music twice a day, each lasting 15 minutes.
  Interventions: Other: the soothing music

INTERVENTIONS:
Other: speech competition training — Speech competition training include voice competition training twice a day in adjunction with drug treatment, and the patients will be required to perform voice-related tasks according to the instruction.
  Arms: a speech competition experimental group
Other: the soothing music — the soothing music
  Arms: Control group

SUMMARY:
One hundred schizophrenia patients with auditory hallucinations will be recruited and randomized into group A and group B. Participants of group A will firstly receive a speech competition training for 2 weeks, and those in group B will firstly receive music intervention as placebo treatment. Specifically, speech competition training include voice competition training twice a day in adjunction with drug treatment, and the patients will be required to perform voice-related tasks according to the instruction. The reaction time, accuracy rate and the number of auditory hallucinations during the task will be recorded. On the other hand, the placebo treatment includes soothing music twice a day for a fixed period of time while patients receiving drug treatment. After 2 weeks, the interventions for group A and group B will be switch.

Clinical symptoms will be evaluated using the auditory hallucinations rating scale, positive and negative syndrome scale, belief about voices questionnaire-revised at baseline, 2-week follow up and 4-week follow up. All the data will be analyzed with the Statistical Product and Service Solutions(SPSS) software.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the diagnostic criteria for schizophrenia as in the International Classification of Diseases (ICD) - 10;
* Aged 18-55 years old;
* Education level over 6 years;
* The score of P3 item in PANSS ≥ 3 points;
* Taking antipsychotics at a therapeutic dose for at least 1 month, and the symptoms of auditory hallucinations have not been significantly improved, and the score of Auditory Hallucinations Rating Scale (AHRS) is still greater than 18 points;
* Capable of understanding and singing a written informed consent form, and be able to cooperate in completing intervention training and assessments.

Exclusion Criteria:

* Diagnosing other Axis I mental disorders;
* A history of severe neurological disease, brain trauma, major physical disease or history of drug dependence;
* Auditory hallucinations caused by organic brain diseases;
* Patients who cannot cooperate with the completion of training;
* Patients with serious suicidal or self injurious behavior;
* Pregnant and lactating women;
* History of alcohol abuse;
* Intellectual impairment (IQ<70);
* Patients with hearing impairment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Auditory Hallucinations Rating Scale (AHRS) | Change of AHRS score from baseline at 2 weeks and 4 weeks respectively
  The Hoffman Hallucination Rating Scale (AHRS) is a clinical tool used to assess the severity of auditory hallucinations in patients. In current study, the scale is used to evaluate the severity of auditory hallucinations in patients with schizophrenia, mainly from seven aspects: frequency, authenticity, loudness, number of sounds, duration, attention significance, and pain level.
Belief About Voices Questionnaire-Revised (BAVQ-R) | Change of BAVQ-R score from baseline at 2 weeks and 4 weeks respectively
  This scale is a self-assessment scale developed by Chadwick et al., used to measure the beliefs, emotions, and behaviors of patients with auditory hallucinations, with a total of 35 items. Straus et al. reconducted factor analysis on its basis and extracted four factors, namely victim belief (authority belief+malicious belief), goodwill belief, participation in auditory hallucinations, and resistance to auditory hallucinations. The scale items are scored using the Likert 4-level scoring method, with a score of 0-3 and independent scores for each dimension.

SECONDARY OUTCOMES:
Negative and Negative Syndrome Scale (PANSS) | Change of PANSS score from baseline at 2 weeks and 4 weeks respectively
  The Negative and Positive Symptoms Scale is a widely used scale for assessing patients' clinical symptoms. The PANSS scale has a total of 30 items, including three subscales of positive symptoms, negative symptoms and general psychopathological symptoms. Each item is scored 1-7 in increasing order of severity. The sum of the items contained in the factor is the factor score, and the scores of all items are added to obtain the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Guo, M.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China